CLINICAL TRIAL: NCT01245166
Title: A Phase III Randomized, Double-blind, Parallel-group Study to Evaluate the Efficacy and Safety of Acarmet (Metformin HCl 500 mg Plus Acarbose 50 mg Tablets) Versus Acarbose Alone in Subjects With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lotus Pharmaceutical (Industry)
Responsible Party: Dr. Wayne-Huey-Herng Sheu, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCCD09013B
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2010-11-22 (Estimated); Status verified 2010-11

CONDITIONS: The Objectives of the Study is to Evaluate the Efficacy and Safety of Acarmet (Metformin HCl 500 mg; Plus Acarbose 50 mg Tablets) Thrice Daily Versus Acarbose 50 mg Thrice Daily Over 16 Weeks in; Subjects With Type 2 Diabetes Mellitus.
MeSH Terms: interventions — Acarbose; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acarbose (Active Comparator)
  Interventions: Drug: Acarbose
- Metformin/Acarbose (Experimental)
  Interventions: Drug: Metformin/Acarbose

INTERVENTIONS:
Drug: Acarbose — Acarbose 50 mg, per orem, thrice daily
  Arms: Acarbose
Drug: Metformin/Acarbose — Metformin HCl 500 mg plus Acarbose 50 mg Tablets, per orem, thrice daily
  Arms: Metformin/Acarbose

SUMMARY:
Type 2 diabetes mellitus is a chronic metabolic disorder which is caused by both insulin secretion deficiency and insulin action defect. In this type of subjects, fasting hyperglycemia is the result of the elevated rate of basal hepatic glucose production, and it is coexisting with hyperinsulinemia.After a meal, the impaired control of hepatic glucose production by insulin and decreased insulin-mediated glucose uptake by muscle contributed nearly equally to postprandial hyperglycemia(Scheen, 1997). Type 2 diabetic subjects experience significant morbidity and mortality from microvascular (retinopathy, nephropathy, and neuropathy) and macrovascular (cardiovascular disease, stroke, and peripheral vascular disease) complications. The appropriate treatment and good glycemic control of diabetes is therefore important and necessary (Vaag, 2006). Evidences suggest that combination therapy using oral antidiabetic agents with different mechanisms of action may be more effective in achieving and maintaining target blood glucose level (Turner et al., 2005).There are five classes of oral antihyperglycemic agents (sulfonylureas, biguanides, α- ucosidase inhibitors, thiazolidinediones and meglitinides) currently available to improve glycemic control in subjects with type 2 diabetes, each of which works through a different mechanism of action. Metformin, a biguanide which has insulin-sensitizing properties, can be used alone or in combination with other classes of agents. Metformin is the currently the first-choice treatment in subjects with diagnosed type 2 diabetic subjects and obesity, characterized by insulin-resistance. Metformin also provides reduction of body weight and ameliorates lipid abnormalities and is thought to be related to a reduction in hepatic gluconeogenesis (Hundal & Inzucchi, 2003).Acarbose, the α-glucosidase inhibitor, is approved for the treatment of type 2 diabetes, and first approved for prediabetes treatment (Chiasson et al., 1994; Breuer, 2003; Chiasson et al., 2002). The drug was launched worldwide as a type 2 diabetes monotherapy and combination therapy in 1990 which has proven efficacious as first-line therapy (Coniff et al., 1995) and in combination with sulfonylureas or insulin (Kelley et al., 1998). Acarbose and metformin are both associated with beneficial effects on hyperglycemia, hyperinsulinemia, body weight, and, in some studies,triglyceride levels (Krentz et al., 1994). Because these factors are part of a cluster of risk factors for cardiovascular disease, combining the two drugs may be useful. In long-term clinical studies, acarbose has shown a favorable safety profile (Hasche et al., 1999).In combination with metformin, acarbose has been shown to improve long-term glycemic control (Rosenstock et al., 1998; Halimi et al., 2000). This study was conducted as a further vestigation into the efficacy and safety of concurrent use of acarbose and metformin in type 2 diabetes mellitus subjects.Lotus Pharmaceutical Co., Ltd. intends to initiate Phase III program to investigate assess the efficacy and safety of metformin in combination with acarbose for type 2 diabetes mellitus subjects considered inadequately blood glucose control. Since combination tablet of acarbose and metformin has not yet been approved by the Taiwan DOH, this study is conducted to evaluate the efficacy and safety of combination tablet of acarbose and metformin in the treatment of type 2 diabetes mellitus subjects in Taiwan. Acarbose is chosen as an active-comparator.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be included in the study only if they meet all of the following criteria:

  1. Male or female subjects aged ≥ 20 and ≤ 80 years old;
  2. Subject with type 2 diabetes mellitus;
  3. Subject with documented HbA1c ≥ 7 % and ≤ 10 % within 3 months prior study and at screening;
  4. Body mass index < 35 kg/m2;
  5. Subject is willing and able to comply with study procedures and sign informed consent.

Exclusion Criteria:

* Subjects will be excluded from the study for any of the following reasons:

  1. Subject with type 1 diabetes or secondary diabetes;
  2. Subject with history or concurrent ketonuria or other acidosis;
  3. Subject with type 2 diabetes mellitus treated with high dose of sulfonylurea (gliclazide > 320 mg, glibenclamide > 20 mg, glimepiride > 6 mg, and glipizide > 20 mg) or with biguanides (metformin > 2000 mg), or of α-glucosidase inhibitors (acarbose > 300 mg), or with meglitinides (repaglinide > 6 mg and nateglinide > 360 mg), thiazolidinedione (rosiglitazone > 4 mg, pioglitazone > 30 mg) or with insulin;
  4. Subject with gastrointestinal disease that may interfere with absorption of the investigational products at discretion of investigator, including but are not limited to malabsorption syndromes and gastric ulcer;
  5. Subject with kidney function impairment defined as serum creatinine > 1.5 mg/dL for male, serum creatinine > 1.4 mg/dL for female, or liver function impairment defined as ALT > 3 X ULN, or AST > 3 X ULN;
  6. Subject with history of drug or alcohol abuse within the past 1 year;
  7. Subject who have been diagnosed with acute myocardial infarction or cardiac failure within 6 months preceding screening;
  8. Subject with hypersensitivity to acarbose and/or metformin products;
  9. Subject with active cancer, defined as ongoing, progressing cancer, or < 5 years of stable disease;
  10. Hemoglobin values < 10 gm/dl for females or <11 gm/dl for males;
  11. Female subject of childbearing potential who:

      * is lactating; or · has positive urine pregnancy test at Visit 1; or
      * refuse to adopt reliable method of contraception during the study;
  12. Subject is contraindicated to acarbose and/or metformin treatment;
  13. Subject has received any investigational agent within 28 days prior to the first dose of investigational product;
  14. Subject who have a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event during the course of the trial, including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine,immune, neurological, or hematological disease as determined by the clinical judgment of the investigator.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The changes from baseline in HbA1c to the end of treatment period | -4 weeks, 0 week, 8 weeks, 12 weeks, 16 weeks

SECONDARY OUTCOMES:
the change from baseline to the end of treatment in FBG, PBG, lipid profiles, and body weight. The safety evaluation will include: 1) Adverse events; 2) Laboratory data; 3) Physical examination; 4) Vital signs; 5) 12- lead ECG | -4 weeks, 0 week, 4 weeks, 8 weeks, 12 weeks, 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan

REFERENCES:
- [Derived] El-Damanawi R, Stanley IK, Staatz C, Pascoe EM, Craig JC, Johnson DW, Mallett AJ, Hawley CM, Milanzi E, Hiemstra TF, Viecelli AK. Metformin for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2024 Jun 4;6(6):CD013414. doi: 10.1002/14651858.CD013414.pub2. PMID 38837240
- [Derived] Wang JS, Huang CN, Hung YJ, Kwok CF, Sun JH, Pei D, Yang CY, Chen CC, Lin CL, Sheu WH; acarbose/metformin fixed-dose combination study investigators. Acarbose plus metformin fixed-dose combination outperforms acarbose monotherapy for type 2 diabetes. Diabetes Res Clin Pract. 2013 Oct;102(1):16-24. doi: 10.1016/j.diabres.2013.08.001. Epub 2013 Aug 15. PMID 23993469